CLINICAL TRIAL: NCT03518021
Title: NTNU Intranasal Naloxone Trial - a Double Blinded, Double Dummy, Randomized Controlled Trial of Intranasal Naloxone for Pre-hospital Use
Brief Title: Naloxone Nasal Spray Compared With Naloxone Injection for Opioid Overdoses Outside the Hospital
Acronym: NINA-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-004072-22; 2016/2000 (Other: REK); 2016-004072-22 (EudraCT Number)
Record Dates: First submitted 2018-05-03; First posted 2018-05-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Overdose; Drug Abuse
Keywords: Naloxone; Administration, Intranasal; Injections, Intramuscular; Narcotic Antagonists
MeSH Terms: conditions — Drug Overdose; Substance-Related Disorders | interventions — Naloxone; Injections, Intramuscular

STUDY DESIGN:
Intervention Model Description: Double blinded, double dummy, randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The whole study team, including the statistician, will be blinded until after database lock and the primary analysis are done. The allocation list will be stored by by the Hospital Pharmacy Trondheim. There will not be automatic unblinding of SAEs. Study personnel do not have any access to the allocation list. An emergency option for individual unblinding is available to medical monitor in case of SAE/ SUSAR Study workers are blinded to the different preparations. This is carefully performed by covering the vials with neutral and opaque labels for "study drug". The risk of for unintentional unblinding is very small. The procedure for securing credible blinding is described in the study protocol and approved by the Norwegian Medicines Agency.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Naloxone, intranasal (Experimental)
  Interventions: Drug: Naloxone, intranasal
- Naloxone, intramuscular (Active Comparator)
  Interventions: Drug: Naloxone, intramuscular
- placebo, intranasal (Placebo Comparator)
  Interventions: Drug: placebo, intranasal
- placebo, intramuscular (Placebo Comparator)
  Interventions: Drug: placebo, intramuscular

INTERVENTIONS:
Drug: Naloxone, intranasal — Active compound naloxone 14 mg/ml, (±10%). Nasal spray will be administered with one puff (100 microL ±10%) in one nostril (1.4 mg dose) using the Aptar Unitdose device.
  The spray device should be inserted about 1 cm into a nostril, pointing towards the ipsilateral ear and the plunger pushed in a firm and gentle manner for the formulation to be sprayed into the nose. After the plunger is inserted the device is immediately removed from the nose and assisted ventilation continued.
  Arms: Naloxone, intranasal
Drug: placebo, intranasal — Same spray but without naloxone. Nasal spray will be administered with one puff (100 microL +/- 10%) in one nostril using the Aptar Unitdose device.
  The spray device should be inserted about 1 cm into a nostril, pointing towards the ipsilateral ear and the plunger pushed in a firm and gentle manner for the formulation to be sprayed into the nose. After the plunger is inserted the device is immediately removed from the nose and assisted ventilation continued.
  Arms: placebo, intranasal
Drug: Naloxone, intramuscular — Intramuscular comparator Naloxone Hydrochloride 0.4 mg/ml will be administered as a 2 ml intramuscular (IM) injection in the deltoid muscle, total dose of 0,8 mg naloxone IM
  Arms: Naloxone, intramuscular
Drug: placebo, intramuscular — Intramuscular Sodium Chloride Injection 9mg/ml, will be administered as a 2 ml intramuscular injection in the deltoid muscle
  Arms: placebo, intramuscular

SUMMARY:
This trial will compare the clinical response to intramuscular and intranasal naloxone in pre-hospital opioid overdoses. Objective of the study is to measure and evaluate clinical response (return of spontaneous respiration within 10 minutes of naloxone administration) to a new nasal naloxone formulation in real opioid overdoses in the pre-hospital environment. The aim is to demonstrate that intranasal administration of naloxone is not clinically inferior to intramuscular administration, which is now standard treatment of care.

ELIGIBILITY:
Inclusion Criteria:

* Suspected opioid overdose clinically diagnosed by emergency medical service (EMS) based on the following criteria

  1. Reduced (below and equal to 8 breaths per minute) or absent spontaneous respiration
  2. Miosis
  3. Glasgow Coma Scale (GCS) below 12
* Palpable carotid or radial arterial pulse

Exclusion Criteria:

* Cardiac arrest
* Failure to assist ventilation using mask-bag technique
* Facial trauma or epistaxis or visible nasal blockage
* Iatrogenic opioid overdose when opioid is administered in- hospital, or by EMS or other health care workers in the pre- hospital setting
* Suspected or visibly pregnant participant
* Has received naloxone by any route in the current overdose
* in prison or custody by police
* EMS staff without training as study workers
* No study drug available
* Study drug frozen as indicated by Freeze Watch in kit or past its expiry date
* Deemed unfit for inclusion due to any other cause by study personnel at the scene; such as unsafe work environment for EMS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with return of spontaneous respiration (above or equal to 10 breaths per minute) within 10 minutes of naloxone administration in pre-hospital opioid overdose | 40 minutes

SECONDARY OUTCOMES:
Changes in Glasgow Coma Scale (GCS) in patients treated with study medicine for opioid overdose | The time participants are in the care of ambulance personnel, estimated 40 minutes
Changes in oxygen saturation (SaO2) in patients treated with study medicine for opioid overdose | The time participants are in the care of ambulance personnel, estimated 40 minutes
Overdose complications | The time participants are in the care of ambulance personnel, estimated 40 minutes
  aspiration, cardiac arrest, death
Time from administration of naloxone to respiration above or equal to 10 breaths per minute | The time participants are in the care of ambulance personnel, estimated 40 minutes
Opioid withdrawal reaction to naloxone reversal | The time participants are in the care of ambulance personnel, estimated 40 minutes
Suitability of spray device in pre-hospital setting | The time participants are in the care of ambulance personnel, estimated 40 minutes
Adverse reactions to naloxone formulation | The time participants are in the care of ambulance personnel, estimated 40 minutes
Need for rescue naloxone, dose and route of administration during study visit | The time participants are in the care of ambulance personnel, estimated 40 minutes
Recurrence of opioid overdose/ need for further pre-hospital naloxone within 12 hours of inclusion | 12 hours
reasons not to give rescue naloxone to non-responders | The time participants are in the care of ambulance personnel, estimated 40 minutes
follow-up after care | The time participants are in the care of ambulance personnel, estimated 40 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, Study Director — Norwegian University of Science and Technology; Arne K Skulberg, MD PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - Oslo University Hospital, Prehospital devision, Oslo
  - St Olavs Hospital, Department for Emergency Medicine and Prehospital Services, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
NTNU has complete ownership and publishing rights of all results, regardless of outcome. The full protocol, Statistical Analysis Plan, information letter for consent and other trial documents will be published open access in the NTNU Open repository. The Clinical Study report and Statistical Analysis Report will also be made openly available, but open versions may be censored to ensure that it will not be possible to identify individual study participants. The datasets analysed during the current study will be made available from NTNU upon reasonable request and a methodological sound proposal based on the consent given by participants.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Updated regularly, but no later than one year after publication of main results
Access Criteria: NTNU will require data processor agreements for recipients conform to standards set out in Norwegian Law and the European General Data Protection Regulation. Any shared datasets will have pseudonymisation of personal data. If doubt NTNU will seek advice from Ethics Committee.
URL: https://dataverse.no/dataset.xhtml?persistentId=doi:10.18710/ABRUWW

REFERENCES:
- [Derived] Skulberg AK, Tylleskar I, Valberg M, Braarud AC, Dale J, Heyerdahl F, Skalhegg T, Barstein J, Mellesmo S, Dale O. Comparison of intranasal and intramuscular naloxone in opioid overdoses managed by ambulance staff: a double-dummy, randomised, controlled trial. Addiction. 2022 Jun;117(6):1658-1667. doi: 10.1111/add.15806. Epub 2022 Feb 8. PMID 35137493
- [Derived] Skulberg AK, Tylleskar I, Braarud AC, Dale J, Heyerdahl F, Mellesmo S, Valberg M, Dale O. NTNU intranasal naloxone trial (NINA-1) study protocol for a double-blind, double-dummy, non-inferiority randomised controlled trial comparing intranasal 1.4 mg to intramuscular 0.8 mg naloxone for prehospital use. BMJ Open. 2020 Nov 12;10(11):e041556. doi: 10.1136/bmjopen-2020-041556. PMID 33184084